CLINICAL TRIAL: NCT03678025
Title: Phase III Randomized Trial of Standard Systemic Therapy (SST) Versus Standard Systemic Therapy Plus Definitive Treatment (Surgery or Radiation) of the Primary Tumor in Metastatic Prostate Cancer
Brief Title: Standard Systemic Therapy With or Without Definitive Treatment in Treating Participants With Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1802; NCI-2018-01738 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1802 (Other: SWOG); S1802 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Castration Levels of Testosterone; Metastatic Prostatic Adenocarcinoma; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abiraterone; bicalutamide; acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Docetaxel; Flutamide; Salicylic Acid; Goserelin; histrelin; Leuprolide; luprolide acetate gel depot; nilutamide; Orchiectomy; Castration; Prednisone; deltacortene; prednylidene; Radiotherapy; Radiation; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Arm I (SST) (Active Comparator): Participants receive 1 acceptable form of SST as in Induction except for treatment with docetaxel and prednisone.
  Interventions: Drug: Abiraterone; Drug: Bicalutamide; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Histrelin Acetate; Drug: Leuprolide Acetate; Drug: Nilutamide; Procedure: Orchiectomy; Other: Quality-of-Life Assessment; Drug: Triptorelin
- Arm II (SST, prostatectomy or radiation therapy) (Experimental): Participants receive 1 acceptable form of SST as in Induction except for treatment with docetaxel and prednisone. Participants undergo prostatectomy within 8 weeks after randomization or radiation therapy within 4 weeks of randomization.
  Interventions: Drug: Abiraterone; Drug: Bicalutamide; Drug: Degarelix; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Histrelin Acetate; Drug: Leuprolide Acetate; Drug: Nilutamide; Procedure: Orchiectomy; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy; Procedure: Radical Prostatectomy; Drug: Triptorelin
- Step 1 (pre-randomization) (Active Comparator): Standard treatment data collection prior to randomization
  Interventions: Drug: Abiraterone; Drug: Bicalutamide; Drug: Degarelix; Drug: Docetaxel; Drug: Flutamide; Drug: Goserelin Acetate; Drug: Histrelin Acetate; Drug: Leuprolide Acetate; Drug: Nilutamide; Procedure: Orchiectomy; Drug: Prednisone; Other: Quality-of-Life Assessment; Drug: Triptorelin

INTERVENTIONS:
Drug: Abiraterone — Given PO
  Other Names: CB 7598
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
Drug: Degarelix — Given via injection
  Other Names: FE200486; Firmagon
Drug: Docetaxel — intravenous
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
  Arms: Step 1 (pre-randomization)
Drug: Flutamide — Given PO
  Other Names: 4'-Nitro-3'-trifluoromethylisobutyranilide; Apimid; Cebatrol; Chimax; Cytomid; Drogenil; Euflex; Eulexine; Flucinom; Flucinome; Flugerel; Fluken; Flulem; FLUT; Fluta-Gry; Flutabene; Flutacan; Flutamex; Flutamin; Flutan; Flutaplex; Fugerel; Grisetin; Niftolide; Oncosal; Profamid; Propanamide, 2-Methyl-N-(4-nitro-3-(trifluoromethyl)phenyl)-; Prostacur; Prostadirex; Prostica; Prostogenat; SCH 13521; Tafenil; Tecnoflut; Testotard
Drug: Goserelin Acetate — Given SC
  Other Names: ZDX; Zoladex
Drug: Histrelin Acetate — Receive SC
  Other Names: Supprelin; Vantas
Drug: Leuprolide Acetate — Receive SC or IM
  Other Names: A-43818; Abbott 43818; Abbott-43818; Carcinil; Depo-Eligard; Eligard; Enanton; Enantone; Enantone-Gyn; Ginecrin; LEUP; Leuplin; Leuprorelin Acetate; Lucrin; Lucrin Depot; Lupron; Lupron Depot; Lupron Depot-3 Month; Lupron Depot-4 Month; Lupron Depot-Ped; Procren; Procrin; Prostap; TAP-144; Trenantone; Uno-Enantone; Viadur
Drug: Nilutamide — Given PO
  Other Names: Anandron; Nilandron; RU-23908
Procedure: Orchiectomy — Undergo bilateral orchiectomy
  Other Names: Castration; Male Castration; Male Gonadectomy; orchidectomy
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
  Arms: Step 1 (pre-randomization)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Standard radiation
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation
  Arms: Arm II (SST, prostatectomy or radiation therapy)
Procedure: Radical Prostatectomy — Standard surgery
  Other Names: Prostatovesiculectomy
  Arms: Arm II (SST, prostatectomy or radiation therapy)
Drug: Triptorelin — injection
  Other Names: 6-D-Tryptophan-LH-RH; 6-D-Tryptophanluteinizing Hormone-releasing Factor; AY-25650; CL-118,532; Decapeptyl; Detryptoreline

SUMMARY:
This phase III trial studies how well standard systemic therapy with or without definitive treatment (prostate removal surgery or radiation therapy) works in treating participants with prostate cancer that has spread to other places in the body. Addition of prostate removal surgery or radiation therapy to standard systemic therapy for prostate cancer may lower the chance of the cancer growing or spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare overall survival in metastatic prostate cancer patients who are randomized to standard systemic therapy (SST) plus definitive treatment of the primary tumor versus standard systemic therapy alone.

SECONDARY OBJECTIVES:

I. To compare overall survival in metastatic prostate cancer patients who received SST plus surgical excision of the primary tumor versus SST alone in the subset who specify the surgical intent stratification factor.

II. To compare the rate of symptomatic local progression between the treatment arms.

III. To compare progression-free survival (PFS) between the two treatment arms. IV. To compare rates of progression-free survival between arms for the subsets of patients with and without metastasis directed therapy (MDT) to oligometastatic sites.

QUALITY OF LIFE OBJECTIVES:

I. To compare between arms patient-reported urinary function and urinary bother over time (after initiation of SST at 6 months, 1, 2, and 3 years) using the Expanded Prostate Cancer Index Composite (EPIC) and patient-reported pain and physical functioning using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) between patients receiving standard systemic therapy and those receiving systemic therapy and definitive management of the primary prostate cancer.

OTHER OBJECTIVES:

I. To bank tissue and whole blood specimens for future use.

OUTLINE:

INDUCTION: Participants receive 1 of 6 acceptable forms of SST for 22-28 weeks. I. Participants undergo a bilateral orchiectomy. II. Participants receive goserelin acetate subcutaneously (SC) every 28 days or 12 weeks, histrelin acetate SC every 12 months, leuprolide acetate SC or intramuscularly (IM) every 1, 3, 4, or 6 months, and triptorelin every 1, 3, or 6 months.

III. Participants receive goserelin acetate SC every 28 days or 12 weeks, histrelin acetate SC every 12 months, leuprolide acetate SC or IM every 1, 3, 4, or 6 months, and triptorelin every 1, 3, or 6 months. Participants also receive nilutamide orally (PO) daily, flutamide PO every 8 hours, and bicalutamide PO daily.

IV. Participants receive degarelix via injection for 2 doses and then every 28 days.

V. Participants receive nilutamide PO daily, flutamide PO every 8 hours, and bicalutamide PO daily. Participants also receive docetaxel over 1 hour every 3 weeks with or without prednisone PO every 12 hours.

VI. Participants receive nilutamide PO daily, flutamide PO every 8 hours, and bicalutamide PO daily. Participants also receive abiraterone PO daily or prednisone PO every 12 hours.

After completion of 22-28 weeks of SST, participants are then randomized to 1 of 2 arms.

ARM I: Participants receive 1 acceptable form of SST as in Induction except for treatment with docetaxel and prednisone.

ARM II: Participants receive 1 acceptable form of SST as in Induction except for treatment with docetaxel and prednisone. Participants undergo prostatectomy within 8 weeks after randomization or radiation therapy within 4 weeks of randomization.

After completion of study treatment, participants are followed up for 8 years.

ELIGIBILITY:
Inclusion Criteria:

* STEP 1 REGISTRATION: DISEASE-RELATED CRITERIA: All patients must have a histologically or cytologically proven diagnosis of adenocarcinoma of the prostate. Patients with pure small cell carcinoma* (SCC), sarcomatoid, or squamous cell carcinoma are not eligible. (*morphology must be consistent with SCC; synaptophysin or chromogranin positive by immunohistochemical staining is insufficient to diagnose SCC).
* STEP 1 REGISTRATION: DISEASE-RELATED CRITERIA: Patients must have an intact prostate. No prior local therapy for prostate adenocarcinoma is allowed (e.g., brachytherapy, high-intensity focused ultrasound [HIFU], cryotherapy, laser ablative therapies). Any prior therapy for benign conditions, such as obstruction, are acceptable (e.g., transurethral resection of the prostate, greenlight laser ablation, microwave ablation).
* STEP 1 REGISTRATION: DISEASE-RELATED CRITERIA: Patients must have evidence of metastatic disease on technetium bone scan and computed tomography (CT) or magnetic resonance imaging (MRI) within 42 days prior to starting standard systemic therapy. Metastatic disease that is detected by positron emission tomography (PET) scan only (sodium fluoride [NaF], prostate-specific membrane antigen [PSMA], anti-1-amino-3-18F-fluorocyclobutane-1-carboxylic acid [FACBC], carbon [C]11) but not conventional imaging (technetium [Tc]99 bone scan, CT or MRI) or solitary metastases by conventional imaging, must be confirmed histologically or cytologically.
* STEP 1 REGISTRATION: DISEASE-RELATED CRITERIA: Patients with known brain metastases are not eligible. Brain imaging studies are not required for eligibility if the patient has no neurologic signs or symptoms suggestive of brain metastasis. If brain imaging studies are performed, they must be negative for disease.
* STEP 1 REGISTRATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients must have received no more than 28 weeks of standard systemic therapy (SST). SST is defined as current National Comprehensive Cancer Network (NCCN) guidelines for metastatic prostate cancer.
* STEP 1 REGISTRATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients must not have progressed while on SST.
* STEP 1 REGISTRATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients with oligometastatic prostate cancer may receive metastasis directed therapy to up to four sites of disease prior to randomization.
* STEP 1 REGISTRATION: CLINICAL/LABORATORY CRITERIA: Patients must have a complete physical examination and medical history within 28 days prior to registration.
* STEP 1 REGISTRATION: CLINICAL/LABORATORY CRITERIA: Patients must have a PSA documented prior to initiation of SST and within 28 days prior to registration. Any additional PSAs measured while receiving SST should be recorded.
* STEP 1 REGISTRATION: CLINICAL/LABORATORY CRITERIA: Patients must have a testosterone lab documented within 28 days prior to randomization. Any additional testosterone labs measured while receiving SST should be recorded as well as pretreatment initiation if available.
* STEP 1 REGISTRATION: CLINICAL/LABORATORY CRITERIA: No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, adequately treated stage 0, I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years.
* STEP 1 REGISTRATION: SPECIMEN SUBMISSION CRITERIA: Patients must be offered the opportunity to participate in translational medicine studies and specimen banking for future studies.
* STEP 1 REGISTRATION: QUALITY OF LIFE CRITERIA: Patients who can complete Patient-Reported Outcome instruments in English, Spanish or French, must participate in the quality of life studies.
* STEP 1 REGISTRATION: REGULATORY CRITERIA: Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* STEP 2 RANDOMIZATION: DISEASE-RELATED CRITERIA: As a part of the OPEN registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.
* STEP 2 RANDOMIZATION: DISEASE-RELATED CRITERIA: Patients must have no evidence of disease progression during the 28 weeks of SST by PSA measure, bone scan and CT or MRI or symptomatic deterioration (as defined by physician discretion) within 28 days prior to randomization.
* STEP 2 RANDOMIZATION: DISEASE-RELATED CRITERIA: Patients must have consultation with a urologist and have surgically resectable disease regardless of definitive treatment intent or randomization.
* STEP 2 RANDOMIZATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients must have received between 22 and 28 weeks of SST as measured from the date of first hormonal therapy or surgical castration. SST is defined by current NCCN guidelines for metastatic prostate cancer.
* STEP 2 RANDOMIZATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients must not be planning to receive docetaxel after randomization.
* STEP 2 RANDOMIZATION: PRIOR/CONCURRENT THERAPY CRITERIA: Any toxicities from SST must have resolved to =< grade 1 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) prior to randomization.
* STEP 2 RANDOMIZATION: PRIOR/CONCURRENT THERAPY CRITERIA: Patients may have received elective metastasis directed therapy to oligometastatic sites (=< 4 sites). All treatment must be completed prior to randomization.
* STEP 2 RANDOMIZATION: CLINICAL/LABORATORY CRITERIA: Patients must have a PSA performed within 28 days prior to randomization.
* STEP 2 RANDOMIZATION: CLINICAL/LABORATORY CRITERIA: Patients must have a testosterone < 50 ng/dL within 28 days prior to randomization.
* STEP 2 RANDOMIZATION: CLINICAL/LABORATORY CRITERIA: Patients must have a Zubrod performance status of 0 ? 1 within 28 days prior to randomization.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1273 (Estimated)
Dates: Start 2018-09-24 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2031-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From date of randomization to date of death due to any cause, assessed up to 8 years

SECONDARY OUTCOMES:
Media OS | From date of randomization to date of death due to any cause, assessed up to 8 years
  Will compare OS in metastatic prostate cancer patients who received standard systemic therapy (SST) plus surgical excision of the primary tumor versus SST alone in the subset who specify the surgical intent stratification factor.
Rate of symptomatic local progression | Up to 8 years
  Defined as any of the following events post-randomization: Common Terminology Criteria for Adverse Events version 5 grade >= 2 hematuria, urinary retention, urinary tract obstruction, urinary tract pain, pelvic pain, renal and urinary disorders-other. Will be compared between the treatment arms. A proportional hazards model will be fit to each of these endpoints where the time interval starts at date of randomization to (i) time of first symptomatic local progression or ii) progression or death due to any cause, where those without the event are censored at their last contact date. Stratification factors will be adjusted for as covariates.
Progression-free survival (PFS) | From date of randomization to date of first documentation of progression, or death due to any cause, assessed up to 8 years
  Will be compared between for the subsets of patients with and without metastasis directed therapy (MDT) to oligometastatic sites. A proportional hazards model will be fit to each of these endpoints where the time interval starts at date of randomization to (i) time of first symptomatic local progression or ii) progression or death due to any cause, where those without the event are censored at their last contact date. Stratification factors will be adjusted for as covariates.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chapin, Principal Investigator — SWOG Cancer Research Network
Locations (338):
- United States (334):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Community Cancer Institute, Clovis, California
  - University Oncology Associates, Clovis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Yale University, New Haven, Connecticut
  - Stamford Hospital/Bennett Cancer Center, Stamford, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Reid Health, Richmond, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Maine Medical Center-Bramhall Campus, Portland, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth/SMHC Cancer Care and Blood Disorders-Sanford, Sanford, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - GenesisCare USA - Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - GenesisCare USA - Farmington Hills, Farmington Hills, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - GenesisCare USA - Macomb, Macomb, Michigan
  - GenesisCare USA - Madison Heights, Madison Heights, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - GenesisCare USA - Troy, Troy, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Upstate Cancer Center Radiation Oncology at Oneida, Oneida, New York
  - Upstate Cancer Center Radiation Oncology at Oswego, Oswego, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - James J Peters VA Medical Center, The Bronx, New York
  - Atrium Health Stanly/LCI-Albemarle, Albemarle, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - Levine Cancer Institute-Gaston, Gastonia, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson in The Woodlands, Conroe, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern Simmons Cancer Center - RedBird, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Lyndon Baines Johnson General Hospital, Houston, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - MD Anderson League City, League City, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Audie L Murphy VA Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - George E Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont Medical Center, Burlington, Vermont
  - Bon Secours Saint Francis Medical Center, Midlothian, Virginia
  - Bon Secours Cancer Institute at Reynolds Crossing, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - FHCC Overlake, Bellevue, Washington
  - Seattle Cancer Care Alliance at EvergreenHealth, Kirkland, Washington
  - FHCC South Lake Union, Seattle, Washington
  - FHCC at Northwest Hospital, Seattle, Washington
  - University of Washington Medical Center - Montlake, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Zablocki Veterans Administration Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Drexel Town Square Health Center, Oak Creek, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- Instituto Nacional del Cancer, Independence, Chile
- Instituto Nacional De Cancerologia, Bogotá, Colombia
- Instituto Nacional De Cancerologia de Mexico, Mexico City, Tlalpan, Mexico
- Kantonsspital Aarau, Aarau, Switzerland